CLINICAL TRIAL: NCT03599037
Title: Use of the ICOUGH RECOVERY App to Improve Protocol Adherence and Post-Operative Outcomes in the Inpatient Space
Brief Title: Inpatient ICOUGH RECOVERY App Version 2.0
Acronym: ICOUGH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators decided not to start up the study after the long Covid 19 pause dring which no participants were enrolled.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-37554
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Post Operative Complications; Pneumonia
Keywords: ICOUGH Recovery App; Length of stay; Care coach; Incentive spirometry; Coughing; Post operative ambulation; Deep breathing; Smartphone
MeSH Terms: conditions — Pneumonia; Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICOUGH Recovery App (Experimental): The ICOUGH Recovery app v2.0 will be downloaded to participants who have a smartphone and want to use the app after their surgery. These participants will be instructed to use the app daily after their surgery until discharge and to select a care coach. Prior to discharge subjects will complete a questionnaire to assess usability and will participate in a brief recorded interview of their experience using the app. Inpatient post operative complications will be abstracted from medical records.
  Interventions: Other: ICOUGH Recovery App v2.0
- Standard of care (No Intervention): Participants who either do not have a smartphone or have a smartphone but don't want to use the app will receive the standard of care after surgery which includes an ICOUGH protocol checklist. Inpatient post operative complications will be abstracted from medical records.

INTERVENTIONS:
Other: ICOUGH Recovery App v2.0 — The app has pre-set auditory, visual reminders, in the form of push notifications, that remind participants to use the incentive spirometer and ambulate around the hospital at time intervals recommended by the ICOUGH protocol. The app benchmarks the level of adherence to that of other subjects involved in the study via the "My Summary" page, and this visual anonymous comparison further motivates adherence to the ICOUGH protocol.
  Arms: ICOUGH Recovery App

SUMMARY:
This pilot study will evaluate how well version 2 of the ICOUGH app, a bed-side mobile app increases patients' adherence to a postoperative protocol called ICOUGH. Specific outcomes, such as length of hospital stay, postoperative lung complications, unplanned intubations, and death will be assessed in participants who do and those who do not use the ICOUGH Recovery app, positing that a smartphone intervention should improve these outcomes over time.

ICOUGH is a mnemonic that stands for each step of a protocol shown to decrease lung-related complications of surgery. It stands for Incentive spirometry (a breathing device that expands the lungs), Coughing and deep breathing, Oral hygiene, Understanding (patient and family education), Getting out of bed at least three times daily, and Head-of-bed elevation.

The ICOUGH protocol was developed at Boston Medical Center (BMC) and has been shown to improve patient outcomes by decreasing postoperative pneumonia by 38%, unplanned intubations by 40%, and all adverse outcomes by 40%, which has resulted in over $5 million in cost savings for BMC in a two-year period. There is an instructional paper pamphlet with intuitive pictures for each step of ICOUGH, and patient subjects can log how many times they've done each step.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility of and adherence to all parts of version 2 of the ICOUGH app, incorporating user feedback and repairing "bugs" discovered during the previous trial. It will also compare postoperative complications and length of stay in participants who used and those who did not use the ICOUGH app. Eligible participants who have a smartphone will decide whether they want to download and use the ICOUGH app or not. Those who choose not to use the app and participants who do not have a smartphone, will receive the postoperative standard of care ICOUGH pamphlet which lists the activities that patients are encouraged to do following surgery to prevent lung complications.

The app incorporates a number of functionalities that encourage subject accountability to the ICOUGH protocol. The participant will be given the option to choose one person from his/her smartphone contact list (friend or family member) to be his/her "care coach." The care coach will first receive an initial text regarding the role of a care coach, which is to help the subject adhere to the ICOUGH protocol. Should the care coach accept this role, he/she will also receive text message updates on the subject's level of adherence to the ICOUGH protocol three times during the day. The care coach is encouraged to help the subject comply with the treatment plan, which he/she can easily do through texting, phone calls, and hospital visits. The patient will be informed of the role and expectations for a care coach during their initial pre-operative assessment clinic visit, prior to consenting. The app will not transmit any private data pertaining to the selected care coach (e.g., name, phone number, etc.) to the back-end server. The concept and function of a care coach is unique to the app and is not ordinarily part of the standard of care.

The app also has pre-set auditory, visual reminders-in the form of push notifications-that remind the subject to use the incentive spirometer and ambulate around the hospital at time intervals recommended by the ICOUGH protocol. Every time the subject interacts with the app, whether by touching its push notifications or interacting with a tablet computer at the nursing station, these interactions can be visualized on the main screen via an intuitive dashboard. Lastly, the app conveniently benchmarks the subject's level of adherence to that of other subjects involved in the study via the "My Summary" page, and this visual comparison is meant to be a form of friendly competition against other (anonymous) patients to further motivate adherence to the protocol.

Following discharge, the research team will perform a retrospective chart review to record participants' length of stay (LOS), development of postoperative pulmonary complications, and other objective data. for participants used and those who did not use the ICOUGH Recovery app.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing emergent general surgery with the Acute Care Surgery service
* English speaker with the ability to read English at 5th grade level
* Able to ambulate, with or without assistance

Exclusion Criteria:

* Presence of neuromuscular disease or inability to perform all the measures in the ICOUGH protocol
* Visually impaired or blind
* Homeless
* Prisoner
* Pregnancy
* Body mass index < 15 kg/m-2 or > 54 kg/m-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Adherence to incentive spirometry | 8 months
  Post operative daily incentive spirometry rates will be calculated from the ICOUGH Recovery app database for those participants who use the app.
Adherence to oral health | 8 months
  Post operative daily oral care rates for ICOUGH app users will be calculated from the ICOUGH Recovery app database for those participants who use the app.
Adherence to ambulation | 8 months
  Post operative daily ambulation rates for ICOUGH app users will be calculated from the ICOUGH Recovery app database for those participants who use the app.

SECONDARY OUTCOMES:
Length of stay | 8 months
  Length of inpatient stay in days will be abstracted from the participants' medical records.
Postoperative pneumonia | 8 months
  Rate of postoperative pneumonia will be calculated from date abstracted from the participants' medical records.
Unplanned intubation | 8 months
  Rates of unplanned intubation will be calculated from date abstracted from the participants' medical records.
Death | 8 months
  Mortality rates will be calculated from date abstracted from the participants' medical records.

OTHER OUTCOMES:
Usability score | 8 months
  A modified System Usability Scale which is a 10 item questionnaire with Likert-style questions with five responses (0 to 4) that range from 'Strongly Disagree' to 'Strongly Agree' will to be completed by participants who use the ICOUGH app. The participant's scores for each question will be converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. A score above a 68 is considered above average and anything below 68 is below average.

CONTACTS AND LOCATIONS:
Overall Officials: David McAneny, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No